CLINICAL TRIAL: NCT04511845
Title: A Phase I, Open-Label, Multicenter, Dose Escalation and Cohort Expansion Study of SPYK04 as Monotherapy in Patients With Locally Advanced or Metastatic Solid Tumors
Brief Title: A Dose-Escalation Study of SPYK04 in Patients With Locally Advanced or Metastatic Solid Tumors (With Expansion).
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chugai Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPK101JG
Record Dates: First submitted 2020-07-08; First posted 2020-08-13 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Locally Advanced or Metastatic Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose escalation cohort of SPYK04 (Experimental): Patients will receive SPYK04 at escalated dose.
  Interventions: Drug: SPYK04
- Expansion part in NSCLC, ovarian cancer and other solid tumors (Experimental): Patients will receive SPYK04 at the recommended dose.
  Interventions: Drug: SPYK04

INTERVENTIONS:
Drug: SPYK04 — SPYK04 capsule

SUMMARY:
Phase I, open-label, multi-center study

ELIGIBILITY:
Inclusion Criteria:

(Both Part I and Part II)

* Age >= 18 years at time of signing informed consent form
* ECOG performance status of 0 or 1
* Patients with a locally advanced, recurrent, or metastatic solid tumor for which standard therapy either does not exist or has proven ineffective or intolerable

(Part I only)

* Patients with measurable and/or evaluable disease per RECIST v1.1
* Patients with MAPK pathway alterations positive solid tumor (i.e., BRAF, K/N/H-RAS mutations)

(Part II only)

* Patients with measurable disease per RECIST v1.1
* Patients with KRAS mutated NSCLC (NSCLC cohort)
* Patients with KRAS mutated Ovarian Cancer (Ovarian Cancer cohort)
* Patients with RAS mutated solid tumor (Biopsy cohort)

Exclusion Criteria:

(Both Part I and Part II)

* Significant cardiovascular disease, such as New York Heart Association (NYHA) cardiac disease (Class II or greater), unstable angina, or myocardial infarction within the previous 6 months or unstable arrhythmias within the previous 3 months
* Patients with primary central nervous system (CNS) malignancy, untreated CNS metastases requiring any anti-tumor treatment, or active CNS metastases
* Patients with current severe, uncontrolled systemic disease (including, but not limited to, clinically significant cardiovascular disease, pulmonary disease, or renal disease, ongoing or active infection)
* Patients with a history or complication of interstitial lung disease (ILD)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Estimated)
Dates: Start 2020-09-10 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of SPYK04 (Dose limiting toxicities) [Dose escalation] | From first dose until the end of Cycle 1 (approximately 35 days)
  Incidence and nature of DLTs
Safety and tolerability of SPYK04 (Adverse Events) [Dose escalation] | From Cycle 0 Day 1 until 28 days after the last dose of study treatment, assessed up to 42 months (study completion)
  Incidence, nature, and severity of adverse events (AEs) as assessed by the NCI CTCAE v5.0
Safety and tolerability of SPYK04 (Electrocardiograms in triplicate) [Dose escalation] | From first dose until the end of Cycle 1 (approximately 35 days)
  Uncorrected QT interval, QTcF, PR duration, QRS interval and RR interval
Safety and tolerability of SPYK04 (Electrocardiograms in triplicate) [Dose escalation] | From first dose until the end of Cycle 1 (approximately 35 days)
  Heart Rate
Pharmacokinetics of SPYK04 [Dose escalation] | From Cycle 0 Day 1 until 28 days after the last dose of study treatment, assessed up to 42 months (study completion)
  Plasma concentrations of SPYK04
Pharmacokinetics of SPYK04 [Dose escalation] | From Cycle 0 Day 1 until 28 days after the last dose of study treatment, assessed up to 42 months (study completion)
  Maximum plasma concentration (Cmax) of SPYK04
Pharmacokinetics of SPYK04 [Dose escalation] | From Cycle 0 Day 1 until 28 days after the last dose of study treatment, assessed up to 42 months (study completion)
  Time to reach maximum plasma drug concentration (Tmax) of SPYK04
Pharmacokinetics of SPYK04 [Dose escalation] | From Cycle 0 Day 1 until 28 days after the last dose of study treatment, assessed up to 42 months (study completion)
  Area under the concentration versus time curve (AUC) of SPYK04
Preliminary anti-tumor activity of SPYK04 [Cohort expansion] | From screening until disease progression, study discontinuation, withdrawal or death, whichever occurs first, assessed up to 42 months (study completion)
  Objective Response Rate (ORR) is defined as proportion of patients who had a confirmed complete response (CR) or partial response (PR), as determined by the investigator with use of Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1)

SECONDARY OUTCOMES:
Preliminary anti-tumor activity of SPYK04 [Dose escalation] | From screening until disease progression, study discontinuation, withdrawal or death, whichever occurs first, assessed up to 42 months (study completion)
  Objective Response
Safety and tolerability of SPYK04 (AEs) [Cohort expansion] | From Cycle 1 Day 1 until 28 days after the last dose of study treatment, assessed up to 42 months (study completion)
  Incidence, nature, and severity of AEs assessed by the NCI CTCAE v5.0
Preliminary anti-tumor activity of SPYK04 [Cohort expansion] | From screening until disease progression, study discontinuation, withdrawal or death, whichever occurs first, assessed up to 42 months (study completion)
  Disease control rate (DCR) is defined as proportion of patients who had an objective response or stable disease (SD), as determined by the investigator with use of RECIST v1.1
Preliminary anti-tumor activity of SPYK04 [Cohort expansion] | From screening until disease progression, study discontinuation, withdrawal or death, whichever occurs first, assessed up to 42 months (study completion)
  Progression-free survival (PFS) is defined as the time from the first study treatment to the first occurrence of progression as determined by the investigator using RECIST v1.1 or death from any cause, whichever occurs first
Preliminary anti-tumor activity of SPYK04 [Cohort expansion] | From screening until disease progression, study discontinuation, withdrawal or death, whichever occurs first, assessed up to 42 months (study completion)
  Duration of response (DoR) is defined for patients with a CR or PR at the time from the first documented CR or PR to documented disease progression as determined by the investigator with use of RECIST v1.1 or death from any cause, whichever occurs first
Pharmacokinetics of SPYK04 [Cohort expansion] | From Cycle 1 Day 1 until 28 days after the last dose of study treatment, assessed up to 42 months (study completion)
  Plasma concentrations of SPYK04
Pharmacokinetics of SPYK04 [Cohort expansion] | From Cycle 1 Day 1 until 28 days after the last dose of study treatment, assessed up to 42 months (study completion)
  Maximum plasma concentration (Cmax) of SPYK04
Pharmacokinetics of SPYK04 [Cohort expansion] | From Cycle 1 Day 1 until 28 days after the last dose of study treatment, assessed up to 42 months (study completion)
  Time to reach maximum plasma drug concentration (Tmax) of SPYK04
Pharmacokinetics of SPYK04 [Cohort expansion] | From Cycle 1 Day 1 until 28 days after the last dose of study treatment, assessed up to 42 months (study completion)
  Area under the concentration versus time curve (AUC) of SPYK04
Pharmacodynamics of SPYK04 [Cohort expansion] | From screening until the time of partial response or stable disease lasting for more than 4 months, and the time of progressive disease, if possible, an average of 1 year
  Expression level of pMEK and pERK in solid tumor tissues (e.g., baseline archival or biopsy, and on treatment biopsy)

CONTACTS AND LOCATIONS:
Overall Officials: Sponsor Chugai Pharmaceutical Co. Ltd, Study Director — clinical-trials@chugai-pharm.co.jp
Locations (15):
- United States (9):
  - Arizona Oncology, Tucson, Arizona
  - Rocky Mountain Cancer Centers, Lone Tree, Colorado
  - Minnesota Oncology, Minneapolis, Minnesota
  - Rhode Island Hospital, Providence, Rhode Island
  - MD Anderson Cancer Center, Houston, Texas
  - Texas Oncology, Tyler, Texas
  - University of Virginia, Charlottesville, Virginia
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Froedtert Hospital and the Medical College of Wisconsin, Milwaukee, Wisconsin
- Japan (6):
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - Kurume University Hospital, Kurume, Fukuoka
  - National Cancer Center Hospital, Chuo Ku, Tokyo
  - Cancer Institute Hospital of Japanese Foundation for Cancer Research, Koto-Ku, Tokyo
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - Osaka Prefectural Hospital Organization Osaka International Cancer Center, Osaka

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform. For further details on Chugai's Data Sharing Policy and how to request access to related clinical study documents, see here (www.chugai-pharm.co.jp/english/profile/rd/ctds_request.html).